CLINICAL TRIAL: NCT07304882
Title: Comparison of Efficacy of Serratiopeptidase and Escin After Impacted Mandibular Third Molar Surgery: A Randomized Controlled Clinical Trial
Brief Title: A Comparison of Recovery After Impacted Wisdom Tooth Removal
Acronym: CESE-3M
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Science and Technology, Yemen (Other)
Responsible Party: Principal Investigator, Arwa Mohammed Dahak, Principal Investigator, University of Science and Technology, Yemen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1445/0012/UREC/UST; ISRCTN15432618 (Registry Identifier: ISRCTN - The UK's Clinical Study Registry)
Record Dates: First submitted 2025-11-21; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: Impacted Mandibular Third Molar Extraction; Post Operative Complications
Keywords: Serratiopeptidase; Escin; Mandibular third molar surgery; Post operative complications; Trismus; Facial edema; Pain; Triple-blind; RCT; Split-mouth design
MeSH Terms: conditions — Trismus; Pain | interventions — serratiopeptidase; Amoxicillin; Metronidazole; Diclofenac; Escin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Serratiopeptidase (Test 1) (Experimental): This group received conventional medications combined with 10 mg oral serratiopeptidase, administered immediately postoperatively and then thrice daily for five days following the first surgical visit.
  Interventions: Drug: serratiopeptidase
- Conventional medication (Control 1) (Active Comparator): During the second visit (after three weeks), only conventional drugs were given. It was consisted of Amoxicillin 500 mg capsules twice daily, Metronidazole 500 mg tablets three times daily, and Diclofenac sodium 50 mg tablets twice daily.
  Interventions: Drug: Conventional drugs
- Escin (Test 2) (Experimental): This group received conventional medications combined with 20 mg oral escin, administered immediately postoperatively and then thrice daily for five days following the first surgical visit
  Interventions: Drug: Escin
- Conventional medication (Control 2) (Active Comparator): During the second visit (after three weeks), only conventional drugs were given. It was consisted of Amoxicillin 500 mg capsules twice daily, Metronidazole 500 mg tablets three times daily, and Diclofenac sodium 50 mg tablets twice daily.
  Interventions: Drug: Conventional drugs

INTERVENTIONS:
Drug: serratiopeptidase — 10 mg oral serratiopeptidase , Amoxicillin 500 mg, Metronidazole 500 mg, Diclofenac sodium 50 mg
  Other Names: Amoxicillin, Metronidazole, and Diclofenac sodium
  Arms: Serratiopeptidase (Test 1)
Drug: Escin — 20 mg oral escin , Amoxicillin 500 mg, Metronidazole 500 mg, Diclofenac sodium 50 mg
  Other Names: Amoxicillin, Metronidazole, and Diclofenac sodium
  Arms: Escin (Test 2)
Drug: Conventional drugs — Amoxicillin 500 mg, Metronidazole 500 mg, Diclofenac sodium 50 mg
  Other Names: Amoxicillin, Metronidazole, and Diclofenac sodium
  Arms: Conventional medication (Control 1); Conventional medication (Control 2)

SUMMARY:
Justification of the Study There is a high prevalence of impacted third molars, often accompanied by a range of postoperative complications. To the best of the researcher's knowledge, no clinical study to date has directly compared the efficacy of serratiopeptidase and escin in minimizing the most commonly observed postoperative complications following impacted mandibular third molar surgery. This study seeks to address this gap by providing empirical evidence that could contribute to optimizing postoperative care.

Objectives of the Study

Drawing from the background and research questions outlined above, the objectives of this study are divided into general and specific ones, outlined as follows:

General Objective To compare the efficacy of serratiopeptidase and escin, when used as adjuncts to conventional drugs, in reducing postoperative complications (i.e., trismus, facial edema, and pain) following impacted mandibular third molar surgery.

Specific Objectives

The study set the following specific objectives:

1. To evaluate the efficacy of serratiopeptidase, as an adjunct to conventional drugs, in reducing postoperative complications (i.e., trismus, facial edema, and pain) following impacted mandibular third molar surgery.
2. To evaluate the efficacy of escin, as an adjunct to conventional drugs, in reducing postoperative complications (i.e., trismus, facial edema, and pain) following impacted mandibular third molar surgery.

Study Hypotheses The study formulated the following hypotheses

1. Serratiopeptidase, as an adjunct to conventional drugs, provides significantly greater efficacy than conventional drugs alone in reducing postoperative complications (i.e., trismus, facial edema, and pain) following impacted mandibular third molar surgery.
2. Escin, as an adjunct to conventional drugs, provides significantly greater efficacy than conventional drugs alone in reducing postoperative complications (i.e., trismus, facial edema, and pain) following impacted mandibular third molar surgery.
3. There is a statistically significant difference in the efficacy of serratiopeptidase compared to escin in reducing postoperative complications (i.e., trismus, facial edema, and pain) when both are used as adjuncts to conventional drugs following impacted mandibular third molar surgery.

DETAILED DESCRIPTION:
This clinical trial employed a split-mouth design, wherein two different treatments were randomly assigned to opposite halves of each patient's mouth. The study was conducted as a triple-blind randomized trial to minimize bias and enhance scientific rigor. The procedures were carried out by the researcher; however, the operator was blinded to the evaluation data. The evaluator, who had access to patients' symptom responses, remained unaware of which treatment was administered on each side. Likewise, patients were blinded to the treatment or intervention applied to each side of their mouth.

Participants were allocated into two groups, with each patient serving as their own control through the split-mouth approach. On one side, an impacted mandibular third molar was extracted and treated with conventional medications. After a washout period of three weeks, the contralateral molar was extracted and treated with an additional intervention alongside the conventional drugs-either an enzyme or a herbal agent. The groups were defined as follows:

* The first group received conventional medications combined with 10 mg oral serratiopeptidase, administered immediately postoperatively and then thrice daily for five days following the first surgical visit. During the second visit (after three weeks), only conventional drugs were given, or vice versa.
* The second group received conventional medications combined with 20 mg oral escin, administered immediately postoperatively and then thrice daily for five days following the first surgical visit. At the second visit (after three weeks), only conventional drugs were administered, or vice versa.

The conventional medication administered to both groups consisted of Amoxicillin 500 mg capsules twice daily, Metronidazole 500 mg tablets three times daily, and Diclofenac sodium 50 mg tablets twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy.
* Presence of two mandibular third molars indicated for surgical extraction.
* No history of pericoronitis or other signs of inflammation within the past 30 days.

Exclusion Criteria:

* Current use of other medications such as NSAIDs or corticosteroids.
* Known allergy to any drugs administered in this study.
* Pregnancy or breastfeeding.
* History of diabetes or hypertension.
* Previous irradiation to the maxillofacial region.
* Intellectual disability or inability to attend follow-up visits.
* Presence of acute or subacute pericoronitis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-01-04 (Actual)

PRIMARY OUTCOMES:
Facial Edema | Baseline measurements were recorded preoperatively. Measurements were reassessed at specific post-operative intervals: immediately after surgery and on the 2nd, 3rd, and 5th postoperative days.
  Facial edema was assessed using the method described by Schultze-Mosgau et al. (1995) to quantitatively evaluate edema both before and after surgery. Measurements were taken with a flexible measuring scale while the patient maintained a closed-mouth position. Five fixed anatomical landmarks and three baseline reference lines were used for consistency:
  • Fixed points: F1 - Tragus of the ear F2 - Angle of the mandible F3 - Soft tissue pogonion F4 - Corner of the mouth F5 - Lateral canthus of the eye
  • Baseline reference lines: S1 - From tragus of the ear to corner of the mouth (Tr-Com) S2 - From tragus of the ear to soft tissue pogonion (Tr-Pgo) S3 - From lateral canthus of the eye to angle of the mandible (Lc-Gn)
Trismus | Baseline measurements were recorded preoperatively. Measurements were reassessed at specific post-operative intervals: immediately after surgery and on the 2nd, 3rd, and 5th postoperative days.
  Trismus was evaluated by measuring the change in maximum mouth opening before and after the surgical procedure. Using a calibrated ruler, the distance between the incisal edges of the upper and lower central incisors was measured in millimeters
Pain Intensity | Baseline measurements were recorded preoperatively. Measurements were reassessed at specific post-operative intervals: immediately after surgery and on the 2nd, 3rd, and 5th postoperative days.
  Pain intensity was evaluated both pre-operatively and post-operatively using a standardized 10-centimeter visual analogue scale (VAS), as described by Sirintawat et al. (2017). The scale ranged from 0, representing no pain, to 10, indicating the worst imaginable pain. At each assessment interval, patients reported the degree of pain they experienced on the scale, providing a simple yet reliable measure of subjective pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Science and Technology, Sanaa, Sana'a, Yemen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chopra D, Rehan HS, Mehra P, Kakkar AK. A randomized, double-blind, placebo-controlled study comparing the efficacy and safety of paracetamol, serratiopeptidase, ibuprofen and betamethasone using the dental impaction pain model. Int J Oral Maxillofac Surg. 2009 Apr;38(4):350-5. doi: 10.1016/j.ijom.2008.12.013. Epub 2009 Jan 24. PMID 19168326
- [Background] Chappi D M, Suresh KV, Patil MR, Desai R, Tauro DP, Bharani K N S S, Parkar MI, Babaji HV. Comparison of clinical efficacy of methylprednisolone and serratiopeptidase for reduction of postoperative sequelae after lower third molar surgery. J Clin Exp Dent. 2015 Apr 1;7(2):e197-202. doi: 10.4317/jced.51868. eCollection 2015 Apr. PMID 26155332
- [Background] Sannino G, Gigola P, Puttini M, Pera F, Passariello C. Combination therapy including serratiopeptidase improves outcomes of mechanical-antibiotic treatment of periimplantitis. Int J Immunopathol Pharmacol. 2013 Jul-Sep;26(3):825-31. doi: 10.1177/039463201302600332. PMID 24067485
- [Background] Bataineh AB, Batarseh RA. The effect of modified surgical flap design for removal of lower third molars on lingual nerve injury. Clin Oral Investig. 2017 Jul;21(6):2091-2099. doi: 10.1007/s00784-016-1999-5. Epub 2016 Nov 12. PMID 27837346
- [Background] Wang T, Fu F, Zhang L, Han B, Zhu M, Zhang X. Effects of escin on acute inflammation and the immune system in mice. Pharmacol Rep. 2009 Jul-Aug;61(4):697-704. doi: 10.1016/s1734-1140(09)70122-7. PMID 19815952
- [Background] Isola G, Matarese M, Ramaglia L, Iorio-Siciliano V, Cordasco G, Matarese G. Efficacy of a drug composed of herbal extracts on postoperative discomfort after surgical removal of impacted mandibular third molar: a randomized, triple-blind, controlled clinical trial. Clin Oral Investig. 2019 May;23(5):2443-2453. doi: 10.1007/s00784-018-2690-9. Epub 2018 Oct 11. PMID 30311061
- [Background] Pavan R, Jain S, Shraddha, Kumar A. Properties and therapeutic application of bromelain: a review. Biotechnol Res Int. 2012;2012:976203. doi: 10.1155/2012/976203. Epub 2012 Dec 10. PMID 23304525
- [Background] Olmedo-Gaya MV, Manzano-Moreno FJ, Galvez-Mateos R, Gonzalez-Rodriguez MP, Talero-Sevilla C, Vallecillo-Capilla M. Oral pregabalin for postoperative pain relief after third molar extraction: a randomized controlled clinical trial. Clin Oral Investig. 2016 Sep;20(7):1819-26. doi: 10.1007/s00784-015-1657-3. Epub 2015 Nov 18. PMID 26578119
- [Background] Villafuerte-Nuñez AE, Téllez-Anguiano AC, Hernández-Díaz O, Rodríguez-Vera R, Gutiérrez-Gnecchi JA, Salazar-Martínez JL. Facial edema evaluation using digital image processing. Discrete Dynamics in Nature and Society. 2013;2013(1):927843. https://doi.org/10.1155/2013/927843
- [Background] Piecuch JF. What strategies are helpful in the operative management of third molars? J Oral Maxillofac Surg. 2012 Sep;70(9 Suppl 1):S25-32. doi: 10.1016/j.joms.2012.04.027. PMID 22916697
- [Background] Kaplan V, Eroglu CN. Comparison of the Effects of Daily Single-Dose Use of Flurbiprofen, Diclofenac Sodium, and Tenoxicam on Postoperative Pain, Swelling, and Trismus: A Randomized Double-Blind Study. J Oral Maxillofac Surg. 2016 Oct;74(10):1946.e1-6. doi: 10.1016/j.joms.2016.05.015. Epub 2016 May 24. PMID 27311846
- [Background] Brkovic B, Andric M, Calasan D, Milic M, Stepic J, Vucetic M, Brajkovic D, Todorovic L. Efficacy and safety of 1% ropivacaine for postoperative analgesia after lower third molar surgery: a prospective, randomized, double-blinded clinical study. Clin Oral Investig. 2017 Apr;21(3):779-785. doi: 10.1007/s00784-016-1831-2. Epub 2016 Apr 25. PMID 27114091
- [Background] Al-Khateeb TH, Nusair Y. Effect of the proteolytic enzyme serrapeptase on swelling, pain and trismus after surgical extraction of mandibular third molars. Int J Oral Maxillofac Surg. 2008 Mar;37(3):264-8. doi: 10.1016/j.ijom.2007.11.011. Epub 2008 Feb 12. PMID 18272344

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT07304882/Prot_SAP_ICF_000.pdf